CLINICAL TRIAL: NCT06068738
Title: Observational Analysis of the Association of Drug Activity Measured in Viable Tumour Tissues ex Vivo and Clinical Response in Ovarian Cancer: A Basic Research Study
Brief Title: Association of Ex Vivo Drug Response (EVDR) and Clinical Outcome in Ovarian Cancer
Acronym: EXCYTE-1
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to a strategic re-evaluation of the company's overall business and clinical development strategy.
Sponsor: Exscientia AI Limited (Industry)
Collaborators: AGO Research GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AC2202
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen viable cells from ascites/pleural effusion and blood, optionally from solid tumour tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly diagnosed: Newly diagnosed ovarian carcinoma patients presenting with ascites and/or pleural effusions before start of their initial therapy.
  Interventions: Other: Biological sample collection
- Relapsed/refractory: Relapsed/refractory (r/r) ovarian carcinoma patients presenting with ascites before start of their next therapy line (for r/r patients).
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — Collection of ascites, blood and fresh tumour tissues (if available)

SUMMARY:
EXCYTE-1 is a multicentre, prospective observational study to investigate the relationship between ex vivo drug response (EVDR), measured in ovarian tumour-derived samples using high content imaging, and actual patient clinical response.

Patients with newly diagnosed or relapsed/refractory epithelial ovarian carcinoma, that present with malignant effusions (ascites or pleural effusions), will be enrolled in the study before starting their initial or next treatment line.

Enrolled patients will be asked to provide ascites, peripheral blood and fresh tumour tissue if available. Samples will be shipped to the sponsor laboratory and their response to standard of care drugs evaluated ex vivo.

Participants will:

* provide samples during routine clinical procedures
* agree that data about their medical history, diagnosis and health status at the following timepoints are collected: at signature of the consent form, at the time samples are provided, at start of the therapy, upon completion of the therapy, regularly after completion of the therapy

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* Signed informed consent form
* Confirmed diagnosis of ovarian cancer except low grade serous, clear cell and mucinous histology
* Where patients are treatment naïve, patients need to have disease stage FIGO (International Federation of Gynecology and Obstetrics) III or FIGO IV.
* Patient is expected to receive primary chemotherapy/maintenance after initial surgical debulking or a further line of systemic therapy in the relapsed setting according to treatment guidelines
* Feasibility of collecting malignant ascites and/or pleural effusion during either primary debulking surgery or a routine drainage procedure prior to initiation of the first or next line of systemic therapy
* ECOG (Eastern Cooperative Oncology Group) stage 0-2

Exclusion Criteria:

* Previously study participation
* Known or suspected HIV or active Hepatitis B and/or C infection or active COVID-19 infection
* Anticancer treatment or radiation therapy of the region which is to be drained or biopsied within the last 4 weeks
* Patient unfit or not willing to receive any further systemic treatment
* Patient is treated with therapeutics not tested in the assay - with the exception of anti-VEGF (Vascular endothelial growth factor) therapy
* Known pregnancy
* Sample quality criteria are not met (at least 250ml of ascites available, no signes of bacterial superinfection, no additives, at least 1% EpCAM (Epithelial Cell Adhesion Molecule) positive cells, viability at least 60%)

Ages: 18 Years to 125 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll newly diagnosed patients with advanced ovarian cancer (FIGO III and FIGO IV) where ascites can be collected during a routine primary debulking surgery, or patients with relapsed (1st, 2nd and 3rd relapse) ovarian cancer scheduled to undergo routine drainage of malignant ascites.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Association between ex vivo drug response (EVDR) of ascites samples and clinical outcome | From time of diagnosis (sampling) until disease progression or End of Study (EoS), whichever comes first, assessed up to 45 month.
  EVDR will be compared to the clinical outcome, determined based on local practice

SECONDARY OUTCOMES:
Technical success rate | From study start to study end (up to 45 month).
  Percentage of ascites samples meeting inclusion and exclusion criteria that meet the quality criteria as per Exscientia SOPs (Standard Operating Procedures).
Prognostic value of EVDR of ascites samples in PFS (Progression-free survival) prediction | From diagnosis until month 6 (12) or relapse/ EoS, whatever comes first.
  False positive and false negative rate in PFS prediction at 6 and 12 month
Biomarker impact on EVDR and its prognostic value | From study start to study end (up to 45 month).
  Hazard rate associated with established biomarkers and interaction between these markers and EVDR outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Krall, Dr., Study Director — Exscientia GmbH
Locations (4):
- Austria (2):
  - Barmherzige Schwestern Linz, Abteilung Gynäkologie und Geburtshilfe, Linz, Upper Austria
  - Med. Universität Wien - Universitätsklinik für Frauenheilkunde, Vienna
- Germany (2):
  - Evang. Kliniken Essen-Mitte gGmbH, Essen, North Rhine-Westphalia
  - Department für Frauengesundheit/Universitäts-Frauenklinik Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kornauth C, Pemovska T, Vladimer GI, Bayer G, Bergmann M, Eder S, Eichner R, Erl M, Esterbauer H, Exner R, Felsleitner-Hauer V, Forte M, Gaiger A, Geissler K, Greinix HT, Gstottner W, Hacker M, Hartmann BL, Hauswirth AW, Heinemann T, Heintel D, Hoda MA, Hopfinger G, Jaeger U, Kazianka L, Kenner L, Kiesewetter B, Krall N, Krajnik G, Kubicek S, Le T, Lubowitzki S, Mayerhoefer ME, Menschel E, Merkel O, Miura K, Mullauer L, Neumeister P, Noesslinger T, Ocko K, Ohler L, Panny M, Pichler A, Porpaczy E, Prager GW, Raderer M, Ristl R, Ruckser R, Salamon J, Schiefer AI, Schmolke AS, Schwarzinger I, Selzer E, Sillaber C, Skrabs C, Sperr WR, Srndic I, Thalhammer R, Valent P, van der Kouwe E, Vanura K, Vogt S, Waldstein C, Wolf D, Zielinski CC, Zojer N, Simonitsch-Klupp I, Superti-Furga G, Snijder B, Staber PB. Functional Precision Medicine Provides Clinical Benefit in Advanced Aggressive Hematologic Cancers and Identifies Exceptional Responders. Cancer Discov. 2022 Feb;12(2):372-387. doi: 10.1158/2159-8290.CD-21-0538. Epub 2021 Oct 11. PMID 34635570